CLINICAL TRIAL: NCT05972486
Title: MUSE Device to Improve Sleep Quality in Midlife Women
Brief Title: A Study of MUSE Device for Midlife Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Amber L. Klindworth, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-000081
Record Dates: First submitted 2023-07-25; First posted 2023-08-02 (Actual); Results first posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Women's Health; Insomnia; Sleep Disturbance
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Parasomnias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Muse-S headband system for management of sleep disturbances (Experimental): Study participants will receive a new Muse-S headband system at study entry and will be asked to utilize it daily for a minimum of 10 minutes day for a period of 6 months (24 weeks). Three of the seven sessions per week will specifically be asked to be mind meditation.
  Interventions: Device: Muse-S™ headband system

INTERVENTIONS:
Device: Muse-S™ headband system — Clinical grade, headband-style wireless EEG (electroencephalogram is a test used to evaluate the electrical activity in the brain) system and designed to interact with a mobile device (a smartphone or tablet). The device is a soft, stretchy band that fits around the forehead to the back of the head.

SUMMARY:
The purpose of this study is to see if it is feasible for midlife women to wear a brain activity sensing headband (Muse-S) for management of sleep disturbances such as insomnia and sleep disruption

ELIGIBILITY:
Inclusion Criteria:

* Women in the menopause transition or in menopause, based on clinical assessment
* PSQI score > 5, with overall sleep quality rating of "fairly bad" or "very bad".
* Motivation VAS score equal to or greater than 5 with overall motivation rating of on a scale of 0-10 with 0 being not motivated at all and 10 being extremely motivated.
* Access to an iPad, iPhone, or android device.
* Have ability to provide informed consent.

Exclusion Criteria:

* Suspected or untreated obstructive sleep apnea.
* Moderate to severe vasomotor symptoms warranting prescription medication use. The FDA categories for hot flash severity are classified as mild (sensation of heat without sweating), moderate (sensation of heat with sweating, able to continue activity), or severe (sensation of heat with sweating cause cessation of activity).
* Use of hormone therapy or hypnotic agents.
* Use of supplements known to affect sleep.
* A known, active, untreated clinically significant psychiatric condition.
* Use of an investigational drug within 30 days of study enrollment or presence of a known history of any condition or factor judged by the investigator to preclude participation in the study or which might hinder adherence.
* Currently (within the past 3 weeks) been practicing mindfulness training on a weekly/regular basis.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-01-12 (Actual); Study Completion 2025-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amber Klindworth, PA-C, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Muse-S Headband System for Management of Sleep Disturbances: Study participants received a new Muse-S headband system at study entry and were asked to utilize it daily for a minimum of 10 minutes day for a period of 6 months (24 weeks). Three of the seven sessions per week were specifically be asked to be mind meditation.
  Muse-S™ headband system: Clinical grade, headband-style wireless EEG (electroencephalogram is a test used to evaluate the electrical activity in the brain) system and designed to interact with a mobile device (a smartphone or tablet). The device is a soft, stretchy band that fits around the forehead to the back of the head.
Period: Overall Study
Arm/Group | Muse-S Headband System for Management of Sleep Disturbances
Started | 31
Completed | 14
Not Completed | 17
Not completed — Withdrawal by Subject | 17

BASELINE CHARACTERISTICS:
Arm/Group | Muse-S Headband System for Management of Sleep Disturbances
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 29
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Change in Quality of Sleep
Description: Measured using the self-reported Pittsburgh Sleep Quality Index (PSQI) to assess the severity of sleep disturbances. Possible scores range from 0 to 21 with higher scores indicating a worse outcome/more severe symptoms of sleep disturbance.
Time Frame: Baseline, 3 months, 6 months
Population: 4 subjects are not included in the change in quality of sleep from baseline to 6-month or change in quality of sleep from 3 months to 6-months as only 14 subjects completed the study through the 6-month time point.
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Muse-S Headband System for Management of Sleep Disturbances
Number analyzed (Participants) | 18
score on a scale
  Baseline to 3 Months | -3 [-4 to -2]
  Baseline to 6 Months: number analyzed (Participants) | 14
  Baseline to 6 Months | -4 [-9 to -3]
  3 Months to 6 Months: number analyzed (Participants) | 14
  3 Months to 6 Months | -1 [-3 to 0]

2. Primary Outcome: Sleep Impact
Description: Measured using the self-reported ASCQ-Me Sleep Impact Short Form. The 5-item questionnaire used to assess functioning and wellbeing in accordance with sleep. The questions in this assessment tool ask how often they felt sleep impacted specific activities during the the past 7 days. Possible answers include: 5 - never; 4 - rarely; 3 - sometimes; 2 - often, and 1 - always. Possible scores range from 5 to 25, with higher scores indicating a better outcome.
Time Frame: Baseline, 3 months, 6 months
Population: 13 subjects are not included in the sleep impact score at 3 months as only 18 subjects completed the study through the 3-month time point. 17 subjects are not included in the sleep impact score at 6 months as only 14 subjects completed the study through the 6-month time point.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Muse-S Headband System for Management of Sleep Disturbances
Number analyzed (Participants) | 31
score on a scale
  Baseline | 18 [8 to 25]
  3 Months: number analyzed (Participants) | 18
  3 Months | 22 [14 to 25]
  6 Months: number analyzed (Participants) | 14
  6 Months | 23 [14 to 25]

3. Secondary Outcome: Perceived Stress Levels
Description: Measured using the self-reported Perceived Stress Scale (PSS). The 10-item questionnaire measures global perceived stress experienced by the participant over the preceding 30 days. The questions in this assessment tool ask how often the participant felt or thought a certain way during the past month. Possible answers include: 0 - never; 1 - almost never; 2 - sometimes; 3 - fairly often, and 4 - very often. Possible scores range from 0 to 40, with lower scores indicating a better outcome (less stress).
Time Frame: Baseline, 3 months, 6 months
Population: 13 subjects are not included in the perceived stress levels score at 3 months as only 18 subjects completed the study through the 3-month time point. 17 subjects are not included in the perceived stress levels score at 6 months as only 14 subjects completed the study through the 6-month time point.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Muse-S Headband System for Management of Sleep Disturbances
Number analyzed (Participants) | 31
score on a scale
  Baseline | 16 [1 to 27]
  3 Months: number analyzed (Participants) | 18
  3 Months | 12 [2 to 21]
  6 Months: number analyzed (Participants) | 14
  6 Months | 12 [4 to 22]

4. Secondary Outcome: Change in Perceived Anxiety
Description: Measured using the self-reported Generalized Anxiety Disorder Scale (GAD-7). The 7-item questionnaire assess severity of generalized anxiety disorder. Scoring is calculated by assigning scores of 0, 1, 2, and 3 to the response categories, respectively, of "not at all," "several days," "more than half the days," and "nearly every day." Total score for the seven items ranges from 0 to 21 where 0 is no anxiety, 1-4 is minimal anxiety, 5-9 is mild anxiety, 10-14 is moderate anxiety, and 15-21 is severe anxiety. With higher scores indicating more severe anxiety.
Time Frame: Baseline, 3 months, 6 months
Population: 4 subjects are not included in the change in perceived anxiety from baseline to 6-month or change in perceived anxiety from 3 months to 6-months as only 14 subjects completed the study through the 6-month time point
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Muse-S Headband System for Management of Sleep Disturbances
Number analyzed (Participants) | 18
score on a scale
  Baseline to 3 Months | -2 [-3 to -1]
  Baseline to 6 Months: number analyzed (Participants) | 14
  Baseline to 6 Months | -2 [-4 to 0]
  3 Months to 6 Months: number analyzed (Participants) | 14
  3 Months to 6 Months | 0 [-5 to 3]

5. Secondary Outcome: Sexual Function
Description: Measured using the self-reported Female Sexual Function Index (FSFI). The 19-item questionnaire to assess the sexual functioning in women. The questions in this assessment tool ask participants about a specific sexual function within the past 4 weeks on a Likert scale range of 0-5. Total scores range from 2 to 36, with lower scores indicating worse sexual functioning.
Time Frame: Baseline, 3 months, 6 months
Population: Only 14 subjects are included in the FSFI scores at 3 months and 6 months as only 14 subjects returned their questionnaire.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Muse-S Headband System for Management of Sleep Disturbances
Number analyzed (Participants) | 21
score on a scale
  Baseline | 18 [2 to 34]
  3 Months: number analyzed (Participants) | 14
  3 Months | 18 [4 to 34]
  6 Months: number analyzed (Participants) | 14
  6 Months | 21 [3 to 33]

6. Secondary Outcome: Sexual Distress
Description: Measured using the Female Sexual Distress Scale (FSDS-R). The 13-item questionnaire to assess sexually related personal distress over the pas 30 days. The questions in this assessment tool asks how often the participant felt during the past month. Possible answers include: 0 - never; 1 - rarely; 2 - occasionally; 3 - frequently, and 4 - always. Possible scores range from 0 to 60, with higher scores indicating greater level of distress.
Time Frame: Baseline, 3 months, 6 months
Population: 8 subjects are not included in the female sexual distress score at 3 months as only 18 subjects completed the study through the 3-month time point. 12 subjects are not included in the female sexual distress score at 6 months as only 14 subjects completed the study through the 6-month time point.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Muse-S Headband System for Management of Sleep Disturbances
Number analyzed (Participants) | 26
score on a scale
  Baseline | 23.5 [13 to 53]
  3 Months: number analyzed (Participants) | 18
  3 Months | 24 [13 to 50]
  6 Months: number analyzed (Participants) | 14
  6 Months | 18 [12 to 41]

7. Secondary Outcome: Change in Quality of Life
Description: Measured using the self-reported Patient Health Questionnaire (PHQ-9). The 9-item questionnaire used to assess severity of depression. Scoring is calculated by assigning scores of 0, 1, 2, and 3 to the response categories, respectively, of "not at all," "several days," "more than half the days," and "nearly every day." Total score for the seven items ranges from 0 to 27 where 0 is no depression, 1-4 is minimal depression, 5-9 is mild depression, 10-14 is moderate depression, and 15-19 is moderately severe depression and 20-27 severe depression. With higher scores indicating more severe depression.
Time Frame: Baseline, 3 months, 6 months
Population: 4 subjects are not included in the change in quality of life from baseline to 6-month or change in quality of life from 3 months to 6-months as only 14 subjects completed the study through the 6-month time point
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Muse-S Headband System for Management of Sleep Disturbances
Number analyzed (Participants) | 18
score on a scale
  Baseline to 3 Months | -2 [-3 to -1]
  Baseline to 6 Months: number analyzed (Participants) | 14
  Baseline to 6 Months | -2 [-3 to -1]
  3 Months to 6 Months: number analyzed (Participants) | 14
  3 Months to 6 Months | 0 [-3 to 1]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of informed consent through study completion, approximately 6 months.
Arm/Group | Muse-S Headband System for Management of Sleep Disturbances
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-31): https://cdn.clinicaltrials.gov/large-docs/86/NCT05972486/Prot_SAP_000.pdf